CLINICAL TRIAL: NCT01731171
Title: A Double-Blind Placebo-Controlled Trial of a Probiotic Supplement to Prevent Relapse and Improve the Clinical Course After Hospitalization for Mania
Brief Title: Probiotics to Prevent Relapse After Hospitalization for Mania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheppard Pratt Health System (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Faith Dickerson, Head, Stanley Research Program, Sheppard Pratt Health System
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SMRI/SPHS: 2012/1
Record Dates: First submitted 2012-11-15; First posted 2012-11-21 (Estimated); Results first posted 2019-01-07 (Actual); Last update posted 2019-01-07 (Actual); Status verified 2019-01

CONDITIONS: Bipolar Disorder; Schizoaffective Disorder
Keywords: mania; manic episode; mixed episode; bipolar disorder; schizoaffective disorder; probiotics; probiotic supplement; relapse prevention; new mood episode; re-hospitalization
MeSH Terms: conditions — Bipolar Disorder; Psychotic Disorders; Mania

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Probiotic Supplement (Experimental): The probiotic supplement compound will consist of capsules containing approximately 10^8 colony forming units of the probiotic organisms, LactobacillusGG and Bifidobacteria lactis strain Bb12. The capsule, which will be swallowed, is a size 3 opaque, hard, hypromellose capsule. The participant will be asked to take 1 capsule of the probiotic supplement with a meal or with a snack daily for 24 weeks.
  Interventions: Dietary Supplement: Probiotic Supplement
- Inert Compound (Placebo Comparator): The inert compound placebo looks identical to the probiotic supplement, and participants will be instructed to swallow 1 capsule with a meal or with a snack daily for 24 weeks.
  Interventions: Dietary Supplement: Inert Compound

INTERVENTIONS:
Dietary Supplement: Probiotic Supplement — Probiotic Supplement 1 tablet by mouth daily
  Other Names: Probio-Tec
  Arms: Probiotic Supplement
Dietary Supplement: Inert Compound — Probiotic identical placebo 1 tablet by mouth daily
  Arms: Inert Compound

SUMMARY:
The purpose of this study is to determine if taking a probiotic supplement versus a placebo will lower rates of relapse and improve the clinical course among participants who have been hospitalized for mania. Relapse and clinical course are measured by time to re-hospitalizations, new mood episodes, and changes in mood-related symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65
* Capacity for written informed consent
* Currently admitted to a Sheppard Pratt inpatient or day hospital for symptoms of mania
* Primary Axis I diagnosis (DSM-IV) at time of admission of Bipolar I Disorder (single manic episode, most recent episode manic, or most recent episode mixed) OR Schizoaffective Disorder, Bipolar type (manic or mixed state)
* Proficient in the English language
* Available to come to Sheppard Pratt Towson for follow-up visits
* Participated previously in one of our screening studies

Exclusion Criteria:

* Diagnosis of mental retardation
* Symptoms of mania secondary to a general medical condition
* Any clinically significant or unstable medical disorder as determined by the investigators including congestive heart failure, abnormal liver function or disease, renal failure, acute pancreatitis, any diagnosis of cancer undergoing active treatment, HIV infection or other immunodeficiency condition
* History of IV drug use
* Primary diagnosis of substance abuse or dependence according to DSM-IV criteria within the last 3 months, or has a positive drug toxicity screen
* Participated in any investigational drug trial in the past 30 days
* Pregnant or planning to become pregnant during the study period
* Receipt of antibiotic medication within the previous 24 hours (as anaerobic organisms residing in the gastrointestinal tract may be minimally affected by antibiotics)
* Documented celiac disease (as such persons should be on a gluten-free diet as this is the standard care). Of note, we are not limiting the study to individuals with elevated levels of gliadin or casein antibodies as we intend to look at these levels as a predictor of response.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Faith Dickerson, PhD, MPH, Principal Investigator — Sheppard Pratt Health System
Locations (1):
- Sheppard Pratt Health System, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dickerson F, Adamos M, Katsafanas E, Khushalani S, Origoni A, Savage C, Schweinfurth L, Stallings C, Sweeney K, Goga J, Yolken RH. Adjunctive probiotic microorganisms to prevent rehospitalization in patients with acute mania: A randomized controlled trial. Bipolar Disord. 2018 Nov;20(7):614-621. doi: 10.1111/bdi.12652. Epub 2018 Apr 25. PMID 29693757

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Probiotic Supplement | Inert Compound
Started | 33 | 33
Completed | 26 | 26
Not Completed | 7 | 7
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Lost to Follow-up | 3 | 2
Not completed — Moved out of Area | 0 | 2
Not completed — Terminated for Lack of Adherence | 0 | 1
Not completed — Terminated for Safety Reasons | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Probiotic Supplement | Inert Compound | Total
Number analyzed (Participants) | 33 | 33 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (11.7) | 33.3 (13.3) | 35.58 (12.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 18 | 42
  Male | 9 | 15 | 24
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Caucasian | 29 | 21 | 50
  Race: African American | 4 | 6 | 10
  Race: Asian | 0 | 2 | 2
  Race: Other | 0 | 4 | 4
Region of Enrollment [Number; unit: participants]
  United States | 33 | 33 | 66

OUTCOME MEASURES:

1. Primary Outcome: Time to First Rehospitalization
Description: The primary outcome was the time to first psychiatric inpatient rehospitalization.
Time Frame: Weeks 0 - 24 of study participation
Measure: Median (Inter-Quartile Range); unit: Days to first readmission
Arm/Group | Probiotic Supplement | Inert Compound
Number analyzed (Participants) | 33 | 33
Days to first readmission | 168 [134 to 169] | 139 [32 to 168]
Statistical Analysis 1: Comparison: Probiotic Supplement vs Inert Compound; Test type: Other — The effect of treatment was calculated using logistic regression and the Cox proportional hazard function employing age, gender, and race as covariates; p = .029, Regression, Logistic; Cox Proportional Hazard = 0.37 — Values less than one favor adjunctive probiotic treatment, while values higher than one favor the placebo

2. Secondary Outcome: Number of Participants Rehospitalized
Description: This is a count of the participants who had at least one rehospitalization during the study period.
Time Frame: Weeks 0 - 24 of study participation
Measure: Count of Participants; unit: Participants
Arm/Group | Probiotic Supplement | Inert Compound
Number analyzed (Participants) | 33 | 33
Participants | 8 | 17
Statistical Analysis 1: Comparison: Probiotic Supplement vs Inert Compound; Test type: Superiority; p = .022, Chi-squared

3. Secondary Outcome: Total Number of Rehospitalizations
Description: This is a count of the number of rehospitalizations in each group during the study period.
Time Frame: Weeks 0 - 24 of study participation
Measure: Number; unit: rehospitalizations
Arm/Group | Probiotic Supplement | Inert Compound
Number analyzed (Participants) | 33 | 33
rehospitalizations | 8 | 24
Statistical Analysis 1: Comparison: Probiotic Supplement vs Inert Compound; Test type: Superiority; p = .009, Regression, Linear

4. Secondary Outcome: Mean Days Rehospitalized
Description: This is the mean number of days rehospitalized for participants in each group during the study period.
Time Frame: Weeks 0 - 24 of study participation
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Probiotic Supplement | Inert Compound
Number analyzed (Participants) | 33 | 33
Days | 2.8 (6.3) | 8.3 (12.4)
Statistical Analysis 1: Comparison: Probiotic Supplement vs Inert Compound; Test type: Superiority; p = .017, Kruskal-Wallis

ADVERSE EVENTS:
Time Frame: Adverse event data are presented for the treatment phase (Weeks 0 - 24) of the trial.
Description: The occurrence of adverse events was assessed by asking participants about problems or health changes at all weekly phone calls and in-person study visits every four weeks throughout the 24-week treatment phase. Reported adverse events were categorized by organ system class.
Arm/Group | Probiotic Supplement | Inert Compound
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/33
Serious Adverse Events (participants affected / at risk) | 8/33 | 17/33
Other Adverse Events (participants affected / at risk) | 31/33 | 29/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Probiotic Supplement (N=33) | Inert Compound (N=33)
Psychiatric rehospitalization (Psychiatric disorders) | 8 (8) | 17 (24)
Hospitalization after a fall (Metabolism and nutrition disorders) | 1 (1) | 0 (0) — This single SAE was a hospitalization for a fall due to hyponatremia.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Probiotic Supplement (N=33) | Inert Compound (N=33)
Gastrointestinal Illness/Condition (Gastrointestinal disorders) | 27 | 25
Cardiovascular Illness/Condition (Cardiac disorders) | 2 | 4
Genitourinary Illness/Conition (Renal and urinary disorders) | 2 | 6
Metabolic and/or Endocrine Illness/Condition (Endocrine disorders) | 3 | 0 — Although these are classified as metabolic and/or endocrine illness/condition in the trial, all AEs in this category fell under Endocrine.
Musculoskeletal Illness/Condition (Musculoskeletal and connective tissue disorders) | 11 | 6
Neurological or Sensory Illness/Condition (Nervous system disorders) | 6 | 10
Respiratory Illness/Condition (Respiratory, thoracic and mediastinal disorders) | 17 | 15
Infections (Infections and infestations) | 2 | 2
Dental Illness/Condition (General disorders) | 2 | 3
Dermatological Illness/Condition (Skin and subcutaneous tissue disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No